CLINICAL TRIAL: NCT06004635
Title: Reliability and Sex-Based Variations in Myotonometer Assessment of Thenar Muscle Properties: Implications for Grip Strength
Brief Title: Reliability of Myotonometry in the Assessment of Mechanical Properties of Thenar Muscles
Status: Completed | Type: Observational
Sponsor: Ilke KARA (Other)
Responsible Party: Sponsor-Investigator, Ilke KARA, Co-Principal Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Other Study IDs: BEU-KTS-02
Record Dates: First submitted 2023-07-24; First posted 2023-08-22 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Muscular Tone
Keywords: rehabilitation; biomechanics; assessment; skeletal muscle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to (i) assess the reliability of myotonometer measurements in determining the mechanical properties of thenar muscle in healthy individuals and explore gender-based variations in these properties; (ii) examine the relationship between pinch grip strength and these mechanical properties.

DETAILED DESCRIPTION:
Investigating the mechanical properties of hand muscles using simple applicable methods such as myotonometer can help to evaluate the effectiveness of programs used in hand rehabilitation, optimize the skills of performance-oriented individuals such as athletes and musicians, and create individualized treatment and training programs. In musculoskeletal-related pathologies such as carpal tunnel syndrome, studying the mechanical properties of the thenar muscles may be important to better understand hand grip strength, hand function and mobility. However, the use of myotonometer in the evaluation of the mechanical properties of the thenar muscles requires a reliability study. Accordingly, the aims of our study are: to (i) assess the reliability of myotonometer measurements in determining the mechanical properties of thenar muscle in healthy individuals and explore gender-based variations in these properties; (ii) examine the relationship between pinch grip strength and these mechanical properties.

ELIGIBILITY:
Inclusion criteria:

* being between 18 and 35 years of age
* having normal upper extremity function
* having a Montreal Cognitive Assessment Test (MoCA) score > 26 points

Exclusion criteria:

* any neuromuscular or musculoskeletal disease
* history of upper limb injury
* upper limb surgery within the last 6 months
* body mass index (BMI) > 30 kg/m2.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults between 18-35 years old
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Muscle tone (Hz) | 30 Minutes
  The muscle tone which is a biomechanical property of the forearm muscles will be evaluated with a portable hand-held myotonometer. This myotonometer (MyotonPRO - Tallinn, Estonia) is non-invasive and provides a quantitative assessment of a muscle's biomechanical properties. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph. To determine the feasibility of the MyotonPRO for assessing the muscle tone of forearm muscles measurements will be performed and recorded.
Stiffness (N/m) | 30 Minutes
  The stiffness which is a biomechanical property of the forearm muscles will be evaluated with a portable hand-held myotonometer. This myotonometer (MyotonPRO - Tallinn, Estonia) is non-invasive and provides a quantitative assessment of a muscle's biomechanical properties. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph. To determine the feasibility of the MyotonPRO for assessing the stiffness of forearm muscles measurements will be performed and recorded.
Elasticity (Logarithmic decrement) | 30 Minutes
  The elasticity which is a viscoelastic property of the forearm muscles will be evaluated with a portable hand-held myotonometer. This myotonometer (MyotonPRO - Tallinn, Estonia) is non-invasive and provides a quantitative assessment of a muscle's viscoelastic properties. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph. To determine the feasibility of the MyotonPRO for assessing the stiffness of forearm muscles measurements will be performed and recorded.

SECONDARY OUTCOMES:
Pinch strength | 30 Minutes
  Pinch grip strength will be assessed using a hydraulic pinchmeter (Baseline). Standard procedures recommended by American Society of Hand Therapists (ASHT) will be followed.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saldiran TC, Schleip R, Tanhan A, Ozturk O, Kara I. Quantifying thenar muscle biomechanical properties: Sex-based variations and implications for grip strength. J Hand Ther. 2025 Jul-Sep;38(3):594-604. doi: 10.1016/j.jht.2024.11.009. Epub 2025 Jan 6. PMID 39765426